CLINICAL TRIAL: NCT04001621
Title: Phase II Study of Pyrotinib in Combination With Capecitabine in Patients With Trastuzumab-resistant HER2-positive Advanced Breast Cancer
Brief Title: Pyrotinib in Combination With Capecitabine in Patients With Trastuzumab-resistant HER2-positive Advanced Breast Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Xichun Hu, professor, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HR-BLTN-003
Record Dates: First submitted 2019-06-27; First posted 2019-06-28 (Actual); Last update posted 2022-12-08 (Actual); Status verified 2022-12

CONDITIONS: Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pyrotinib plus capecitabine (Experimental): pyrotinib(400 mg once daily) + capecitabine (2000 mg/m^2 daily, 1000 mg/m^2 BID)
  Interventions: Drug: Pyrotinib combined with capecitabine

INTERVENTIONS:
Drug: Pyrotinib combined with capecitabine — pyrotinib 400 mg once daily; Capecitabine 1000 mg/m2 per day on day 1 through 14, every 21 days.

SUMMARY:
Trastuzumab resistance, which is a common therapeutic challenge in HER2 positive metastatic breast cancer, is not fully understood. Pyrotinib is an oral tyrosine kinase inhibitor targeting EGFR, HER-2 and HER-4 receptors. More general inhibition of ErbB family with pyrotinib could provide additional benefit. This study is designed to evaluate the efficacy and safety of pyrotinib in combination with capecitabine in patients with HER2 positive locally advanced or metastatic breast cancer who had early failure on or after trastuzumab treatment.

DETAILED DESCRIPTION:
A multi-center, one-arm, open label design study, which is planned to enroll 100 patients with trastuzumab-resistant HER2-positive advanced breast cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Pathologically confirmed HER2 positive patients with locally advanced or metastatic breast cancer: HER2 IHC 3+, or HER2 IHC 2+ and FISH detection gene amplification
2. Aged ≥18 and ≤70 years.
3. ECOG performance status of 0 to 1.
4. Life expectancy of more than 12 weeks;
5. At least one measurable lesion exists(RECIST 1.1)
6. Patients with trastuzumab resistance is defined as follows:

   Progression during or within 12 months after treatment in neoadjuvant or adjuvant setting (at least 9 weeks of trastuzumab treatment); Or Progression during or within 6 months after treatment for locally advanced or metastatic disease in the first-line setting (at least 6 weeks of trastuzumab treatment).
7. At least 4 weeks from the last treatment of trastuzumab or chemotherapy，at least 5 times of t1/2 or 4 weeks from the last treatment of endocrine therapy（the shorter one is preferred）
8. Known hormone receptor status
9. For patients with brain metastases, local treatment (including whole cranial radiotherapy, SBRT, etc.) is required and the brain lesions are stable for ≥ 3 months without the need for dexamethasone or mannitol treatment
10. Patients with adequate organ function before enrollment:

    1. ANC≥1.5×10^9/L
    2. PLT≥100×10^9/L
    3. Hb≥90 g/L
    4. TBIL≤1.5×ULN
    5. ALT and AST≤3×ULN, （ALT and AST≤5×ULN in patients with liver metastases）
    6. Cr≤1.5×ULN and the creatinine clearance rate≥50 mL/min
    7. LVEF ≥ 50%
    8. QTcF < 480 ms
11. Signed informed consent.

Exclusion Criteria:

1. Patients with meningeal metastasis and / or spinal cord metastasis;
2. Patients unable to swallow, with chronic diarrhea, intestinal obstruction, or multiple factors that affect drug use and absorption;
3. Patients with malignant serious effusion which cannot be controlled by drainage or other methods;
4. Less than 4 weeks from the last treatment in last clinical trial;
5. Known dihydropyrimidine dehydrogenase (DPD) deficiency;
6. Receiving any other antitumor therapy;
7. History of other malignancy within the last 5 years, except for carcinoma in situ of cervix, basal cell carcinoma or squamous cell carcinoma of the skin that has been previously treated with curative intent;
8. Received radiotherapy, surgery (excluding local puncture) within 4 weeks prior to enrollment; received anti-tumor endocrine therapy after entering the screening period;
9. Previous or ongoing use of HER2-targeted tyrosine kinase inhibitors (lapatinib, neratinib or pyrotinib);
10. Previous use of capecitabine or capecitabine not tolerated, except that capecitabine efficacy cannot be judged or capecitabine discontinuation for 3 months or more;
11. Patients with serious heart disease;
12. Allergy to pyrotinib; history of immunodeficiency, including HIV positive, active HBV/HCV or other acquired, congenital immunodeficiency disease, or organ transplantation history;
13. Known history of neurological or psychiatric disease, including epilepsy or dementia;
14. Patients during pregnancy or lactation, patients with childbearing potential tested positive in baseline pregnancy test, or patients unwilling to take effective contraceptive measures throughout the trial;
15. Evidence of significant medical illness that will substantially increase the risk on the participation or completion of the study in the investigator's judgment. Examples included, but not limited to, hypertension, severe diabetes, etc;
16. Patients not eligible for this study judged by the investigator.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-06-26 (Actual); Primary Completion 2023-05-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) | Estimated 12 months
  From enrollment to progression or death (for any reason)

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | Estimated 12 months
  Ratio of CR and PR in all subjects
Duration of Response (DOR) | Estimated 12 months
  The first evaluation of CR or PR to progression or death (for any reason)
Clinical Benefit rate (CBR) | Estimated 12 months
  Ratio of CR,PR and SD greater than or equal to 24 weeks in all subjects
Overall Survival (OS) | Estimated 24 months
  From enrollment to death (for any reason)
Adverse Events and Serious Adverse Events | From informed consent through 28 days following treatment completion
  Safety

CONTACTS AND LOCATIONS:
Overall Officials: Xichun Hu, Principal Investigator — Department of Oncology
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, China

REFERENCES:
- [Derived] Cao J, Teng Y, Li H, Zhang L, Ouyang Q, Xie W, Pan Y, Song Z, Ling X, Wu X, Xu J, Li L, Ren L, Wang H, Zhou D, Luo J, Hu X. Pyrotinib plus capecitabine for trastuzumab-resistant, HER2-positive advanced breast cancer (PICTURE): a single-arm, multicenter phase 2 trial. BMC Med. 2023 Aug 9;21(1):300. doi: 10.1186/s12916-023-02999-0. PMID 37559142